CLINICAL TRIAL: NCT01181206
Title: Standard-Bauchwandabdeckung Mit Bauchtüchern vs. Abdeckung Mittels ringförmiger Folie: Eine Doppelblinde Randomisiert-kontrollierte Studie
Brief Title: Covering of the Abdominal Wall in Laparotomies: Differences in Surgical Site Infections Between an Approved Abdominal 3M™ Steri-Drape™ Wound Edge Protector and Standard Woven Swabs at Technische Universität München
Acronym: BaFo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TUM-Chir-002/2010
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2012-12

CONDITIONS: Comparing the Number of Surgical Site Infections; Covering of the Abdominal Wall in Laparotomies With an Approved Abdominal 3M™ Steri-Drape™ Wound Edge Protector and Standard Woven; Swabs
Keywords: Surgical site infections; Covering the abdominal wound edge in laparotomies
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Procedure: Intervention Arm 1: Covering with approved abdominal 3M™ Steri-Drape™ Wound Edge Protector Intervention Arm 2: Covering with standard woven swabs
- Arm 2 (Active Comparator)
  Interventions: Procedure: Intervention Arm 1: Covering with approved abdominal 3M™ Steri-Drape™ Wound Edge Protector Intervention Arm 2: Covering with standard woven swabs

INTERVENTIONS:
Procedure: Intervention Arm 1: Covering with approved abdominal 3M™ Steri-Drape™ Wound Edge Protector Intervention Arm 2: Covering with standard woven swabs

SUMMARY:
BaFo is a prospective, double-blinded randomized controlled clinical trial that assesses the numbers of surgical site infections in two different techniques of covering the abdominal wall in laparotomies. Standard covering with woven swabs is compared to a novel, approved 3M™ Steri-Drape™ Wound Edge Protector.

ELIGIBILITY:
Inclusion Criteria:

* Ability to sign the informed consent
* Patients older than 18 years
* Abdominal operations with longitudinal / cross section with clean wounds, clean-contaminated wounds or contaminated wounds (cdc-definitions of surgical wound infections)

Exclusion Criteria:

* Pregnant or lactating women
* Revision Operations
* Operations with dirty or infected wounds (CDC definition of surgical wound infections)
* Laparoscopic operations
* Small operations without longitudinal- / cross-section e.g. appendectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Surgical site infections | 3 years

SECONDARY OUTCOMES:
Body-Temperature during Operation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Friess, M.D., Principal Investigator — Department of Surgery, Klinikum rechts der Isar der Technischen Universität München; Joerg Kleeff, M.D., Principal Investigator — Department of Surgery, Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Department of Surgery and Institute of Statistics Klinikum rechts der Isar der Technischen Universität München, München, Bavaria, Germany

REFERENCES:
- [Derived] Mihaljevic AL, Schirren R, Ozer M, Ottl S, Grun S, Michalski CW, Erkan M, Jager C, Reiser-Erkan C, Kehl V, Schuster T, Roder J, Clauer U, Orlitsch C, Hoffmann TF, Lange R, Harzenetter T, Steiner P, Michalski M, Henkel K, Stadler J, Pistorius GA, Jahn A, Obermaier R, Unger R, Strunk R, Willeke F, Vogelsang H, Halve B, Dietl KH, Hilgenstock H, Meyer A, Kramling HJ, Wagner M, Schoenberg MH, Zeller F, Schmidt J, Friess H, Kleeff J. Multicenter double-blinded randomized controlled trial of standard abdominal wound edge protection with surgical dressings versus coverage with a sterile circular polyethylene drape for prevention of surgical site infections: a CHIR-Net trial (BaFO; NCT01181206). Ann Surg. 2014 Nov;260(5):730-7; discussion 737-9. doi: 10.1097/SLA.0000000000000954. PMID 25379844
- [Derived] Mihaljevic AL, Michalski CW, Erkan M, Reiser-Erkan C, Jager C, Schuster T, Schuhmacher C, Kleeff J, Friess H. Standard abdominal wound edge protection with surgical dressings vs coverage with a sterile circular polyethylene drape for prevention of surgical site infections (BaFO): study protocol for a randomized controlled trial. Trials. 2012 May 15;13:57. doi: 10.1186/1745-6215-13-57. PMID 22587425